CLINICAL TRIAL: NCT02329847
Title: A Phase 1/2a Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of the Combination of Ibrutinib With Nivolumab in Subjects With Hematologic Malignancies
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of the Combination of Ibrutinib With Nivolumab in Participants With Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR106681; PCI-32765LYM1002 (Other: Janssen Research & Development, LLC); 2014-005191-28 (EudraCT Number)
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Neoplasms
Keywords: Hematologic Neoplasms; JNJ54179060; Ibrutinib; Nivolumab
MeSH Terms: conditions — Hematologic Neoplasms | interventions — ibrutinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (6):
- Cohort A1 (Experimental): Participants will receive ibrutinib 420 milligram (mg) capsule orally once daily and nivolumab intravenously as 3 milligram/kilogram (mg/kg) every 2 weeks for 14-daily dosing cycles and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Nivolumab
- Cohort A2 (Experimental): Participants will receive ibrutinib 560 mg capsule orally once daily and nivolumab intravenously as 3 mg/kg every 2 weeks for 14-daily dosing cycles and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Nivolumab
- Cohort B1 (Experimental): Participants will receive ibrutinib recommended Phase 2 dose (RP2D) orally once daily and nivolumab intravenously as 3 mg/kg every 2 weeks for 14-daily dosing cycles and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Nivolumab
- Cohort B2 (Experimental): Participants will receive ibrutinib recommended Phase 2 dose (RP2D) orally once daily and nivolumab intravenously as 3 mg/kg every 2 weeks for 14-daily dosing cycles and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Nivolumab
- Cohort B3 (Experimental): Participants will receive ibrutinib recommended Phase 2 dose (RP2D) orally once daily and nivolumab intravenously as 3 mg/kg every 2 weeks for 14-daily dosing cycles and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Nivolumab
- Cohort B4 (Experimental): Participants will receive ibrutinib recommended Phase 2 dose (RP2D) orally once daily and nivolumab intravenously as 3 mg/kg every 2 weeks for 14-daily dosing cycles and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib — Participants will receive oral capsule of ibrutinib once daily as either 420 mg or 560 mg or at recommended Phase 2 dose in any of the cohort.
  Other Names: JNJ54179060
Drug: Nivolumab — Participants will receive nivolumab intravenously as 3 mg/kg on Day 1 every cycle of 14 days.
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to determine the safety and to establish the recommended phase 2 dose (RP2D) for the combination of ibrutinib and nivolumab in participants with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), follicular cell lymphoma (FL) and diffuse large B-cell lymphoma (DLBCL). Once the dose is optimized, the combination will be assessed for Pharmacokinetics, Pharmacodynamics, and preliminary efficacy, further safety in participants with CLL/SLL, FL or DLBCL and in participants with Richter syndrome.

DETAILED DESCRIPTION:
This is an open-label study, which consists of Part A (Dose Optimization Cohorts) and Part B (Expansion Cohorts). Part A consists of two dose optimization cohorts (cohort A1 and cohort A2) will determine the RP2D for the combination based on safety, pharmacokinetic, and pharmacodynamic assessments in participants with relapsed/refractory CLL/SLL or B-cell non-Hodgkin lymphoma (B-NHL). Part B consists 3 participant populations to further evaluate the safety and clinical activity of ibrutinib in combination with nivolumab: Cohort B1 (participants with CLL/SLL with del 17p or del 11q), Cohort B2 (participants with FL), Cohort B3 (participants with DLBCL) and Cohort B4 (participants with Richter syndrome). Part A and B will consist of Screening Period (28 days before enrollment), Treatment Period and Follow up Period (every 3 months until death or the end of study). Participants will receive nivolumab intravenously (Day 1 of every cycle) and ibrutinib orally once daily on a 14-day cycle. Efficacy will primarily be evaluated by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) and International Working Group (IWG) for lymphoma guidelines. Participants' safety will be monitored throughout the study. Further exploration of pharmacokinetic/pharmacodynamic and biomarker information will be assessed throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status grade 0, 1, or 2
* Adequate bone marrow, liver, and renal function defined as: 1) Absolute neutrophil count (ANC) greater than equal to (>=) 1.5* 10^9cells/litre (L); 2) Platelets >=75 x 109cells/L without transfusion support within 7 days prior to test; 3) Hemoglobin >= 8 gram/deciliter (g/dL) without transfusion support within 7 days prior to test 4) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than equal to (<=) 2.5 * upper limit of normal (ULN) 5) Total bilirubin less than (<) 2 milligram/deciliter (mg/dL) 6) Creatinine determined by serum creatinine levels <=1.5 * ULN or a calculated creatinine clearance of >= 50 mL/min/1.73 m^2
* Histologically confirmed B-cell non-Hodgkin lymphoma (B-NHL), Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
* Relapsed refractory disease after at least 1 but not more than 4 lines of previous systemic therapy
* Measurable disease (NHL: At least 1 measurable site of disease [>1.5 centimeter [cm] in the long axis regardless of short axis measurement or >1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions])
* Cohort B-1: SLL/CLL: 1) Deletion of short arm of chromosome 17 or 11 q based on institutional assessment 2) Relapsed/refractory after at least 1 prior systemic therapy 3) Active disease based in IWCLL criteria
* Cohort B-2: 1) B- cell follicular lymphoma Grade 1, 2, or 3a (WHO criteria) 2) Relapsed/refractory disease >= 2 lines separated by Progression, prior treatment (or not eligible for receiving) CD20 antibody 3) Measurable disease (IWG -Lugano 2014)
* Cohort B-3: 1) Histologically-confirmed DLBCL 2) Prior standard rituximab + anthracyclin containing regimen, received or not eligible or considered candidate of HD-ASCT 3) Measurable disease (IWG -Lugano 2014)
* Cohort B-4: 1) Histologically-confirmed Richter syndrome defined as transformation of CLL or SLL into an aggressive lymphoma 2) Previously treated with at least one line of standard, systemic chemotherapy or not eligible for standard therapy 3) At least 1 measurable site of disease based on the Revised Response Criteria for Malignant Lymphoma

Exclusion Criteria:

* Prior therapy or surgery (3 to 10 weeks depending type)
* Prior BTK inhibitor or anti PD1, anti PDL1, anti PD-L2 and anti-CD137, anti-cytotoxic T-lymphocyte associated antigen (CTLA-4) antibody
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification, or congenital long QT syndrome, or QT interval corrected for heart rate, using Fridericia formula (QTcF) at Screening greater than (>) 470 milliseconds (ms)
* History of stroke or intracranial hemorrhage within 6 months prior to the first dose of ibrutinib
* Requires treatment with anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong cytochrome P450 3A (CYP3A) inhibitors
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (18):
- New York, New York, United States
- Australia (3):
  - Bedford Park
  - Darlinghurst
  - Woolloongabba
- Israel (4):
  - Haifa
  - Jeursalem
  - Ramat Gan
  - Tel Aviv
- Poland (4):
  - Chorzów
  - Gdansk
  - Krakow
  - Wroclaw
- Spain (3):
  - Barcelona
  - Madrid
  - Salamanca
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir

REFERENCES:
- [Derived] Bruscaggin A, di Bergamo LT, Spina V, Hodkinson B, Forestieri G, Bonfiglio F, Condoluci A, Wu W, Pirosa MC, Faderl MR, Koch R, Schaffer M, Alvarez JD, Fourneau N, Gerber B, Stussi G, Zucca E, Balasubramanian S, Rossi D. Circulating tumor DNA for comprehensive noninvasive monitoring of lymphoma treated with ibrutinib plus nivolumab. Blood Adv. 2021 Nov 23;5(22):4674-4685. doi: 10.1182/bloodadvances.2021004528. PMID 34500472
- [Derived] Younes A, Brody J, Carpio C, Lopez-Guillermo A, Ben-Yehuda D, Ferhanoglu B, Nagler A, Ozcan M, Avivi I, Bosch F, Caballero Barrigon MD, Hellmann A, Kuss B, Ma DDF, Demirkan F, Yagci M, Horowitz NA, Marlton P, Cordoba R, Wrobel T, Buglio D, Streit M, Hodkinson BP, Schaffer M, Alvarez J, Ceulemans R, Balasubramanian S, de Jong J, Wang SS, Fourneau N, Jurczak W. Safety and activity of ibrutinib in combination with nivolumab in patients with relapsed non-Hodgkin lymphoma or chronic lymphocytic leukaemia: a phase 1/2a study. Lancet Haematol. 2019 Feb;6(2):e67-e78. doi: 10.1016/S2352-3026(18)30217-5. Epub 2019 Jan 11. PMID 30642819

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg: Participants with chronic lymphocytic leukemia (CLL)/ follicular cell lymphoma (FL)/diffuse large B-cell lymphoma (DLBCL), received ibrutinib 420 milligrams (mg) capsule orally once daily starting from Day 1 of Cycle 1 up to 56 cycles (26 months). Participants also received nivolumab 3 mg/kilogram (kg) as an intravenous (IV) infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg: Participants with FL/DLBCL, received ibrutinib 560 mg capsule orally once daily starting from Day 1 of Cycle 1 up to 56 cycles (26 months). Participants also received nivolumab 3 mg/kg as an IV infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg: Participants with CLL/small lymphocytic lymphoma (SLL) with deletion (del) 17p or 11q, received ibrutinib 420 mg orally once daily, starting at 7 days prior to Day 1 of Cycle 1 as a run-in period and then daily thereafter up to 56 cycles (26 months). Participants also received nivolumab 3 mg/kg as an IV infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg: Participants with FL, received ibrutinib 560 mg orally once daily, starting at 7 days prior to Day 1 of Cycle 1 as a run-in period and then daily thereafter up to 56 cycles (26 months). Participants also received nivolumab 3 mg/kg as an IV infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg: Participants with DLBCL, received ibrutinib 560 mg orally once daily, starting from Day 1 of Cycle 1 up to 56 cycles (26 months), along with nivolumab 3 mg/kg administered as an IV infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg: Participants with richter syndrome, received ibrutinib 560 mg orally once daily, starting from Day 1 of Cycle 1 up to 56 cycles (26 months), along with nivolumab 3 mg/kg administered as an IV infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
Period: Overall Study
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
Started | 7 | 7 | 36 | 35 | 39 | 20
Treated (Safety Analysis Set) | 7 | 7 | 35 | 35 | 37 | 20
Completed | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 7 | 7 | 35 | 35 | 39 | 20
Not completed — Death | 4 | 4 | 22 | 12 | 20 | 13
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 5 | 7 | 8 | 3
Not completed — Other | 1 | 2 | 6 | 13 | 10 | 3

BASELINE CHARACTERISTICS:
Population: The all-treated population included all participants who had received at least 1 dose of study drugs (either ibrutinib or nivolumab).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Total
Number analyzed (Participants) | 7 | 7 | 35 | 35 | 37 | 20 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (18.08) | 65.9 (13.96) | 64.3 (9.57) | 61.3 (11.94) | 59.2 (15.99) | 64.9 (11.19) | 62.2 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 9 | 15 | 10 | 12 | 54
  Male | 3 | 3 | 26 | 20 | 27 | 8 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 3 | 0 | 0 | 4
  Not Hispanic or Latino | 7 | 7 | 34 | 31 | 35 | 20 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 1 | 2 | 0 | 5
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 5 | 35 | 33 | 34 | 20 | 134
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 0 | 0 | 2 | 1 | 8 | 1 | 12
  ISRAEL | 6 | 1 | 4 | 8 | 6 | 0 | 25
  POLAND | 0 | 0 | 18 | 6 | 6 | 10 | 40
  SPAIN | 1 | 3 | 5 | 6 | 2 | 4 | 21
  TURKEY | 0 | 0 | 6 | 6 | 8 | 1 | 21
  UNITED STATES | 0 | 3 | 0 | 8 | 7 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Assessed International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008: Disease Cohort
Description: ORR is percentage of participants achieving a complete response (CR), CR with incomplete marrow recovery (CRi), nodular partial response (nPR) or PR. IWCLL 2008 criteria: CR- No lymphadenopathy and hepatosplenomegaly, no constitutional symptoms, neutrophils >1.5*10^9/L, platelets >100*10^9/L, Hgb >11 g/dL and absolute lymphocyte count <4000/mcL; CRi- CR with incomplete recovery of bone marrow; nPR- participants meet criteria for CR, but the bone marrow biopsy shows B-lymphoid nodules, may represent a clonal infiltrate; PR- >=50% drop in lymphocyte count from baseline or <=4.0*10^9/L with following: >=50% decrease in sum products of up to 6 lymph nodes, no new enlarged lymph nodes, When abnormal, >=50% decrease in enlargement of spleen from baseline or normalization and a response in 1 of following: Neutrophils >1.5*10^9/L, Platelets>100000/mcL and Hgb>11 g/dL or >=50% improvement over baseline in all. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: Up to 6 years 11 months
Population: The all-treated population included all participants who had received at least 1 dose of study drugs (either ibrutinib or nivolumab). The ORR evaluation criteria were disease specific and hence the analysis was done as per disease cohorts for this outcome measure as pre-planned.
Measure: Number; unit: Percentage of Participants
Groups:
- Ibrutinib and Nivolumab: Chronic Lymphocytic Leukemia (CLL): Participants with CLL in Cohort A1 and B1, received ibrutinib 420 milligrams (mg) capsules orally, daily starting at 7 days prior to Day 1 of Cycle 1 as a run-in period and then daily thereafter up to 56 cycles (26 months). Participants also received nivolumab 3 mg/kilograms (kg) as an intravenous (IV) infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
Arm/Group | Ibrutinib and Nivolumab: Chronic Lymphocytic Leukemia (CLL)
Number analyzed (Participants) | 30
Percentage of Participants | 63.3

2. Primary Outcome: Overall Response Rate (ORR) as Assessed Non-Hodgkin Lymphoma (NHL), Cheson 2014: Disease Cohort
Description: ORR defined as percentage of participants achieving a CR, CRi, nPR or PR. As per Non-Hodgkin Lymphoma, Cheson 2014, CR is complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. PR is >= 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. Progressive disease (PD) >= 50% increase from nadir in the sum of the products of at least two lymph nodes, or appearance of a new lesion greater than 1.5 cm in any axis even if other lesions are decreasing in size. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Up to 6 years 11 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- Ibrutinib and Nivolumab: Small Lymphocytic Lymphoma (SLL): Participants with SLL in Cohort B1, received ibrutinib 420 mg capsules orally, daily starting at 7 days prior to Day 1 of Cycle 1 as a run-in period and then daily thereafter up to 56 cycles (26 months). Participants also received nivolumab 3 mg/kilograms (kg) as an intravenous (IV) infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Ibrutinib and Nivolumab: Follicular Lymphoma (FL): Participants with FL in Cohorts A1, A2, and B2, and who had histologically confirmed initial diagnosis of FL, received ibrutinib either 420 or 560 mg capsules orally, daily starting at 7 days prior to Day 1 of Cycle 1 as a run-in period and then daily thereafter up to 56 cycles (26 months). Participants also received nivolumab 3 mg/kilograms (kg) as an intravenous (IV) infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Ibrutinib and Nivolumab: Diffuse Large B-cell Lymphoma (DLBCL): Participants with DLBCL in Cohorts A1, A2, and B3, and who had histologically confirmed disease with at least 1 measurable disease site, received ibrutinib either 420 or 560 mg capsules orally, daily starting on Day 1 of Cycle 1 up to 56 cycles (26 months), along with nivolumab 3 mg/kg administered as an IV infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
- Ibrutinib and Nivolumab: Richter: Participants who had histologically confirmed Richter syndrome in Cohort B4 with at least 1 site of measurable disease, received ibrutinib 560 mg capsules orally, daily starting on Day 1 of Cycle 1 up to 56 cycles (26 months), along with nivolumab 3 mg/kg administered as an IV infusion on Day 1 of each cycle up to 56 cycles. Each cycle was of 14 days.
Arm/Group | Ibrutinib and Nivolumab: Small Lymphocytic Lymphoma (SLL) | Ibrutinib and Nivolumab: Follicular Lymphoma (FL) | Ibrutinib and Nivolumab: Diffuse Large B-cell Lymphoma (DLBCL) | Ibrutinib and Nivolumab: Richter
Number analyzed (Participants) | 6 | 40 | 45 | 20
Percentage of Participants | 50.0 | 32.5 | 37.8 | 65.0

3. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Event (TEAEs): Study Cohort
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. TEAEs for the treatment phase included events with an onset date/time on or after the start of study intervention through end of study were considered as treatment-emergent.
Time Frame: Up to 6 years 10 months
Population: The safety population included all participants who received at least 1 dose of study drugs (either ibrutinib or nivolumab).
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 7 | 7 | 35 | 35 | 37 | 20
Percentage of Participants | 100 | 100 | 100 | 100 | 97.3 | 95.0

4. Secondary Outcome: Duration of Response (DoR): Study Cohort
Description: DOR is defined as the interval between the date of initial documentation of a response including partial response with lymphocytosis (PRL) and date of first documented evidence of progressive disease or death or date of censoring. iWCLL 2008 criteria for progressive disease: New enlarged nodes >1.5 cm, new hepatomegaly or splenomegaly, or other organ infiltrates; >= 50% increase from nadir in existing lymph node or >=50% increase from nadir in sum of product of diameters of multiple nodes; >=50% increase from nadir in enlargement of liver or spleen; >=50% increase from baseline in lymphocyte count (>=5*10^9/L) unless considered treatment-related lymphocytosis; new cytopenia (Hemoglobin b or platelets) attributable to CLL; transformation to a more aggressive histology.
Time Frame: Up to 6 years 11 months
Population: The all-treated population included all participants who had received at least 1 dose of study drugs (either ibrutinib or nivolumab) and achieved either PR or better (including PRL only for CLL participants).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 2 | 1 | 26 | 12 | 15 | 13
Months | 11.5 [2.4 to 20.7] | NA [NA to NA] — Here 'NA' indicates that median and 95% CI could not be estimated due to less number of participants with events. | 19.2 [9.4 to 19.4] | 10.2 [5.1 to 17.8] | NA [4.6 to NA] — Here 'NA' indicates that median and upper limit of 95% CI could not be estimated due to less number of participants with events. | 6.9 [1.3 to NA] — Here 'NA' indicates that upper limit of 95% CI could not be estimated due to less number of participants with events.

5. Secondary Outcome: Duration of Stable Disease or Better: Study Cohort
Description: Duration of stable disease or better was defined as duration from the start of the treatment until the criteria for progression were met. IWCLL 2008 criteria for progressive disease: New enlarged nodes >1.5 cm, new hepatomegaly or splenomegaly, or other organ infiltrates; >= 50% increase from nadir in existing lymph node or >=50% increase from nadir in sum of product of diameters of multiple nodes; >=50% increase from nadir in enlargement of liver or spleen; >=50% increase from baseline in lymphocyte count (and to >=5*10^9/L) unless considered treatment-related lymphocytosis; new cytopenia (Hemoglobin b or platelets) attributable to CLL; transformation to a more aggressive histology.
Time Frame: Up to 6 years and 11 months
Population: The all-treated population included all participants who had received at least 1 dose of study drugs (either ibrutinib or nivolumab) and met criteria for progressive disease. Here 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 1 | 1 | 5 | 7 | 1 | 0
Months | 24.8 [24.8 to 24.8] | 20.8 [20.8 to 20.8] | 17.38 [14.0 to 21.6] | 14.55 [12.7 to 20.4] | 14.1 [14.1 to 14.1] |

6. Secondary Outcome: Progression-free Survival (PFS): Study Cohort
Description: PFS is defined as the duration from the date of first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death, whichever comes first. Participants who were progression-free and alive or had unknown status were censored at the last tumor assessment. IWCLL 2008 criteria for progressive disease: New enlarged nodes >1.5 cm, new hepatomegaly or splenomegaly, or other organ infiltrates; >= 50% increase from nadir in existing lymph node or >=50% increase from nadir in sum of product of diameters of multiple nodes; >=50% increase from nadir in enlargement of liver or spleen; >=50% increase from baseline in lymphocyte count (and to >=5*10^9/L) unless considered treatment-related lymphocytosis; new cytopenia (Hemoglobin b or platelets) attributable to CLL; transformation to a more aggressive histology.
Time Frame: Up to 6 years 11 months
Population: The all-treated population included all participants who had received at least 1 dose of study drugs (either ibrutinib or nivolumab) and met criteria for progressive disease.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 6 | 5 | 16 | 26 | 22 | 11
Months | 2.0 [1.1 to 24.8] | 9.1 [0.7 to 20.8] | 21.6 [12.0 to 21.6] | 7.6 [2.9 to 12.7] | 3.2 [2.1 to NA] — Here 'NA' indicates that upper limit of 95% CI could not be estimated due to less number of participants with events. | 5.0 [2.4 to NA] — Here 'NA' indicates that upper limit of 95% CI could not be estimated due to less number of participants with events.

7. Secondary Outcome: Overall Survival (OS): Study Cohort
Description: OS was defined as duration from the date of first dose of study drug to the date of the participant's death.
Time Frame: Up to 6 years 11 months
Population: The all-treated population included all participants who had received at least 1 dose of study drugs (either ibrutinib or nivolumab) and were responders.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 4 | 3 | 11 | 9 | 16 | 8
Months | 12.4 [2.0 to 28.8] | NA [0.8 to NA] — Here 'NA' indicates that median and upper limit of 95% CI could not be estimated due to less number of participants with events. | NA [21.6 to NA] — Here 'NA' indicates that median and upper limit of 95% CI could not be estimated due to less number of participants with events. | NA [NA to NA] — Here 'NA' indicates that median and 95% CI could not be estimated due to less number of participants with events. | 19.0 [7.7 to NA] — Here 'NA' indicates that upper limit of 95% CI could not be estimated due to less number of participants with events. | 10.3 [4.8 to NA] — Here 'NA' indicates that upper limit of 95% CI could not be estimated due to less number of participants with events.

8. Secondary Outcome: Percentage of Participants With Lymphoma-related Symptoms: Study Cohort
Description: Percentage of participants with lymphoma-related symptoms were reported. These symptoms included B-symptoms, recurrent fever, night sweats, weight loss, other disease-related symptoms, itching, fatigue, physical discomfort and any other.
Time Frame: Up to 6 years 11 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 7 | 7 | 35 | 35 | 37 | 20
Percentage of Participants | 14.3 | 42.9 | 74.3 | 25.7 | 54.1 | 60.0

ADVERSE EVENTS:
Time Frame: Up to 6 years 11 months
Description: All-cause mortality was assessed on all randomized participants. Serious adverse events and other adverse events were assessed on safety analysis set which included all participants who received at least 1 dose of study drugs (either ibrutinib or nivolumab).
Arm/Group | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 4/7 | 4/7 | 22/36 | 12/35 | 20/39 | 13/20
Serious Adverse Events (participants affected / at risk) | 4/7 | 3/7 | 23/35 | 15/35 | 23/37 | 15/20
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 35/35 | 35/35 | 35/37 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg (N=7) | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=7) | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg (N=35) | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=35) | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=37) | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 3 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cardiotoxicity (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal Compression (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 2 | 1
Unevaluable Event (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Biliary Obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis Media Chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2 | 1 | 2
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia Klebsiella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia Parainfluenzae Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Immunoglobulins Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Transaminases Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Leukaemic Infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Penile Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1 (CLL/FL/DLBCL): Ibrutinib 420 mg + Nivolumab 3 mg/kg (N=7) | Cohort A2 (FL/DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=7) | Cohort B1 (CLL/SLL): Ibrutinib 420 mg + Nivolumab 3 mg/kg (N=35) | Cohort B2 (FL): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=35) | Cohort B3 (DLBCL): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=37) | Cohort B4 (Richter Syndrome): Ibrutinib 560 mg + Nivolumab 3 mg/kg (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 9 | 5 | 11 | 8
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 20 | 7 | 10 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 11 | 5 | 7 | 3
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 3 | 2 | 2 | 1
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 3 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0
Euthyroid Sick Syndrome (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 3 | 1 | 3 | 0
Eye Haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 2 | 0
Lacrimation Increased (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Miosis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 3 | 5 | 5 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 3 | 2 | 1 | 1
Anal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 3 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 13 | 12 | 12 | 5
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3 | 3 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 7 | 9 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 3 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 6 | 1
Asthenia (General disorders) | 1 | 2 | 3 | 5 | 1 | 1
Chills (General disorders) | 1 | 0 | 1 | 2 | 2 | 1
Fatigue (General disorders) | 2 | 3 | 6 | 14 | 11 | 1
Gait Disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Generalised Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 2 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 4 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 0 | 7 | 3 | 3 | 3
Pain (General disorders) | 0 | 1 | 1 | 1 | 1 | 1
Peripheral Swelling (General disorders) | 0 | 1 | 2 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 10 | 5 | 9 | 6
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Secondary Immunodeficiency (Immune system disorders) | 0 | 0 | 2 | 0 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 4 | 2 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 3 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 2 | 2 | 1 | 1 | 2
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus Infection Reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Gallbladder Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 1
Herpes Simplex (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 0
Klebsiella Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 4 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 2
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 3 | 5 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 0
Pulpitis Dental (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 3 | 2 | 0 | 0
Rhinovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 4 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 11 | 10 | 7 | 7
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 3 | 2 | 3 | 2
Viral Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Viral Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Wound Infection Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 0
Nasal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 4 | 4 | 5 | 4
Amylase Increased (Investigations) | 1 | 1 | 5 | 1 | 3 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 4 | 3 | 3 | 4
Blood Alkaline Phosphatase (Investigations) | 0 | 0 | 0 | 1 | 2 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 3 | 1 | 3 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 2 | 1 | 2 | 2
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 2 | 3 | 2 | 5 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Blood Uric Acid Increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0
Lipase Increased (Investigations) | 2 | 2 | 8 | 2 | 5 | 3
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 2 | 1 | 1 | 2
Serum Ferritin Decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
Weight Decreased (Investigations) | 0 | 0 | 2 | 2 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 3 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 8 | 6 | 7 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 5 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 2 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 10 | 5 | 5 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 4 | 5 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 4 | 9 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 3 | 3 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 6 | 3 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 3 | 0
Dizziness Postural (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 5 | 5 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 3 | 3 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 2 | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 2 | 3 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 3 | 2 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4 | 11 | 5 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 4 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 3 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5 | 3 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 | 1 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 6 | 8 | 11 | 4
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3 | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 5 | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 4 | 4 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0 | 2 | 3
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
White Coat Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Though it was planned to administer Ibrutinib 280 milligrams (mg) to participants in case the toxicity increased, no participants received ibrutinib 280 mg in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT02329847/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT02329847/SAP_001.pdf